CLINICAL TRIAL: NCT07098533
Title: Cognicise Training for Seniors for Healthy Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 124/21
Record Dates: First submitted 2025-07-09; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Depressive Symptom; Cognitive Functions; Quality of Life; Physical Fitness; Blood Biomarkers; Elderly (People Aged 65 or More); Postural Stability; Fall Risk; Postmenopausal Women; Cardiopulmonary
Keywords: elderly; yoga; cognicise; women; training; exercise
MeSH Terms: conditions — Depression; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Yoga Group (Experimental): Participants in this group completed 16 yoga sessions over 8 weeks. Sessions were conducted twice a week and lasted 60 minutes each. Each session included a warm-up (15 minutes), a main part (30 minutes), and relaxation exercises (15 minutes). The practice focused on movements for the upper and lower limbs and the torso, especially the lumbar spine, pelvis, and hips. The final 10 minutes of each session were dedicated to achieving a deep relaxation state.
  Interventions: Behavioral: Yoga Training
- Cognicise Group (Experimental): Participants in this group completed 16 Cognicise training sessions over 8 weeks. Sessions were held twice a week and lasted 60 minutes. Each session followed a dual-task format combining motor and cognitive elements. Participants performed basic physical exercises while responding to live piano music and visual color cues. They also completed simple language tasks (e.g., spelling words backwards, naming items in categories) and arithmetic tasks. The session structure included a 15-minute warm-up, 30 minutes of cognitive-motor training, and 15 minutes of relaxation and breathing exercises.
  Interventions: Behavioral: Cognicise Training
- Control Group (No Intervention): Participants in the control group did not participate in any structured physical or cognitive training during the 8-week intervention period. They were instructed to maintain their usual daily routines and not to begin any new exercise or therapy programs. Baseline and post-intervention assessments were conducted at the same time points as in the intervention groups.

INTERVENTIONS:
Behavioral: Cognicise Training — The Cognicise program included 16 sessions over 8 weeks (twice weekly, 60 minutes each). This dual-task training combined motor activities with cognitive exercises. During basic gymnastic movements, participants responded to real-time changes in live music and visual stimuli while also solving simple verbal and math tasks. Sessions were divided into 15 minutes of warm-up, 30 minutes of dual-task activity, and 15 minutes of breathing and relaxation exercises.
  Arms: Cognicise Group
Behavioral: Yoga Training — The yoga intervention consisted of 16 instructor-led sessions over 8 weeks (twice weekly, 60 minutes each). Each session included a warm-up (15 minutes), a main phase (30 minutes) focused on exercises targeting the spine, pelvis, and hips, and a relaxation period (15 minutes), including 10 minutes of deep relaxation techniques.
  Arms: Yoga Group

SUMMARY:
The goal of this clinical trial is to assess the impact of two 8-week motor-cognitive exercise programs - Cognicise and yoga - on psychological, respiratory, cardiovascular, postural, and biochemical health in elderly women.

The main objectives are to evaluate whether these programs:

Improve psychological parameters such as mood, quality of life, depressive symptoms, and cognitive abilities;

Enhance respiratory function, including lung volumes and ventilation;

Influence cardiovascular parameters such as blood pressure and heart rate;

Improve chest mobility, physical fitness, and cardiorespiratory capacity;

Induce favorable changes in selected blood biomarkers, including neurotrophic factors, hormones, glucose, lipids, and blood morphology;

Improve postural stability, as assessed through posturographic analysis.

The study compares the effects of yoga and Cognicise to a control group that does not receive any intervention.

Participants in the yoga and Cognicise groups will take part in supervised sessions twice a week for 8 weeks (each session lasting 45 minutes).

Participants from all three groups (yoga, Cognicise, and control) will undergo pre- and post-intervention assessments, including:

Psychological questionnaires;

Spirometry and cardiorespiratory tests;

Blood pressure and heart rate measurements;

Chest mobility and physical fitness tests;

Posturographic assessment of postural control during quiet standing with eyes open and closed;

Laboratory blood tests (including BDNF, GDNF, 25(OH)D, TSH, testosterone, cortisol, insulin, glucose, lipid profile, and complete blood count with differential).

The aim is to determine whether structured motor-cognitive training leads to measurable health benefits compared to no intervention.

ELIGIBILITY:
Inclusion Criteria:

Women aged over 65 years; Community-dwelling; Score of at least 7 points on the Abbreviated Mental Test Score (AMTS).

Exclusion Criteria (presence of at least one of the following):

Locomotor system disorders preventing independent movement; Morbid obesity; Active or stable cancer (ongoing radiation or chemotherapy); Liver disease with ALT > 3× upper limit of normal; Chronic kidney disease (eGFR < 30 mL/min/1.73 m²); Acute inflammation (CRP > 5 mg/dL); Unstable ischemic heart disease; History of ischemic or hemorrhagic stroke within the last 6 months; History of STEMI with drug-eluting stent implantation; NSTEMI within the past 12 months; Inherited metabolic disorders (e.g., phenylketonuria, galactosemia); Autoimmune diseases (e.g., acute thyroiditis, celiac disease, systemic connective tissue disease, hemolytic anemia, vitiligo, Addison's disease, hyperbilirubinemia); Non-specific enteritis (e.g., Crohn's disease, ulcerative colitis); Psychological disorders; Current antibiotic therapy; Current steroid therapy.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Maximal Oxygen Uptake (VO₂max) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Predicted VO₂max estimated using a modified Åstrand-Ryhming protocol on a cycle ergometer. Higher values indicate better cardiovascular fitness. Units: milliliters per kilogram per minute (mL/kg/min)
Geriatric Depression Scale (GDS) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  GDS-15 (15 items). Scores range from 0 to 15; higher scores indicate more severe depressive symptoms. Units: score (0-15; higher = worse outcome)
Brain-Derived Neurotrophic Factor (BDNF) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Serum concentration of BDNF measured in fasting blood samples collected in the morning. Units: ng/mL.

SECONDARY OUTCOMES:
Rosenberg Self-Esteem Scale | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Stroop test10-item scale. Scores range from 0 to 30; higher scores indicate greater self-esteem. Units: score (0-30; higher = better outcome).
Beck Depression Inventory (BDI-II) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  21-item inventory. Scores range from 0 to 63; higher scores indicate greater depressive symptoms. Units: score (0-63; higher = worse outcome).
Stroop Test - Completion Time | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Time (in seconds) to complete the interference condition of the Stroop Test. Lower values indicate better executive functioning. Units: seconds (s).
Stroop Test - Number of Errors | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Number of errors during the interference condition. Lower scores indicate better cognitive control. Units: count.
Body Mass Index (BMI) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Calculated as body mass (kg) divided by height (m) squared. Units: kg/m².
Fat Mass | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Body fat percentage measured using bioimpedance analysis. Units: %.
Muscle Mass | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Skeletal muscle mass percentage via bioimpedance analysis. Units: %.
Visceral Fat | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Visceral fat level assessed via bioimpedance analysis, expressed as an index score. Units: score.
Chest Expansion | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Thoracic expansion measured with tape during maximum inspiration and expiration. Units: centimeters (cm).
Vital Capacity - Percentage of Predicted | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Vital capacity expressed as a percentage of predicted value based on age, sex, and height. Units: %.
Minute Ventilation (VE) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Volume of air exhaled per minute. Units: liters per minute (L/min).
Tidal Volume (TV) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Volume of air exhaled in one breath. Units: milliliters (mL).
Respiratory Rate (RR) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Number of breaths per minute during resting conditions. Units: breaths per minute (brpm).
FEV1/FVC Ratio | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Ratio of forced expiratory volume in one second to forced vital capacity. Units: percentage (%).
Maximal Expiratory Flow (MEF75, MEF50, MEF25) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Maximal flow at selected points of forced expiration, expressed as a percentage of predicted. Units: percentage (%).
Heart Rate (HR) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Measured at rest using standard heart rate monitor. Units: beats per minute (bpm).
Systolic Blood Pressure (SBP) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Measured in mmHg using standard sphygmomanometer. Units: millimeters of mercury (mmHg).
Diastolic Blood Pressure (DBP) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Measured in mmHg using standard sphygmomanometer. Units: millimeters of mercury (mmHg).
Borg Rating of Perceived Exertion (RPE) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Subjective perception of exertion using a 1-10 scale. Units: score (1-10).
White Blood Cells (WBC) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Measured from fasting serum sample. Units: mg/dL.
Red Blood Cells (RBC) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Total erythrocyte count. Units: 10¹²/L.
Hemoglobin (HGB) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Hemoglobin concentration in blood. Units: g/dL.
Hematocrit (HCT) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Proportion of blood volume occupied by red cells. Units: percentage (%).
Red Cell Distribution Width (RDW-CV) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Coefficient of variation of red blood cell size distribution. Units: percentage (%).
Platelets (PLT) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Platelet count. Units: 10⁹/L.
Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Differential white blood cell count. Units: percentage (%).
Total Cholesterol (TC) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Measured from fasting serum sample. Units: mg/dL.
HDL Cholesterol (HDL) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  High-density lipoprotein cholesterol. Units: mg/dL.
LDL Cholesterol (LDL) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Low-density lipoprotein cholesterol. Units: mg/dL.
Triglycerides (TG) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Serum triglyceride concentration. Units: mg/dL.
Glucose (GLU) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Fasting glucose concentration. Units: mg/dL.
Thyroid Stimulating Hormone (TSH) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Serum TSH level. Units: μIU/mL.
Insulin (INS) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Serum insulin concentration. Units: μIU/mL.
Cortisol (COR) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Morning serum cortisol level. Units: µg/dL.
Testosterone (TES) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Total serum testosterone concentration. Units: ng/mL.
Testosterone to Cortisol Ratio (T/C) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Ratio of serum testosterone to cortisol. Units: unitless (arbitrary units).
Glial Cell Line-Derived Neurotrophic Factor (GDNF) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Serum concentration of GDNF. Units: ng/mL.
Irisin (IRS) | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Serum irisin concentration. Units: ng/mL.
Posturography - Displacements of Center of Pressure - Path Length: | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program)
  Total path length of center of pressure displacement during quiet standing. Units: mm.
Posturography - Displacements of Center of Pressure - the total area enclosed by the COP trajectory | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program).
  Assessment of postural stability during quiet standing for 30 seconds with eyes open and eyes closed. Measurement of the total area enclosed by the COP trajectory in square centimeters (cm²).
Posturography - Center of Pressure Path Length to its Area enclosed ratio | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program).
  Assessment of postural stability during quiet standing for 30 seconds with eyes open and eyes closed. Ratio of COP path length to the enclosed area (unitless).
Posturography - Displacements of Center of Pressure - average Speed | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program).
  Assessment of postural stability during quiet standing for 30 seconds with eyes open and eyes closed. Average speed of COP displacement measured in centimeters per second (cm/s).
Posturography - Displacements of Center of Pressure - average x-axis speed | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program).
  Assessment of postural stability during quiet standing for 30 seconds with eyes open and eyes closed. Average speed of COP displacement along the x-axis in centimeters per second (cm/s).
Posturography - Displacements of Center of Pressure - average y-axis speed | Baseline (within 3 days before intervention) and Post-intervention (within 3 days after the 8-week program).
  Assessment of postural stability during quiet standing for 30 seconds with eyes open and eyes closed. Average speed of COP displacement along the y-axis in centimeters per second (cm/s).

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Gronek, Prof., Study Chair — Poznan University of Physical Education
Locations (1):
- Poznan University of Physical Education, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Yes